CLINICAL TRIAL: NCT00523549
Title: A Multi-center, Prospective, Randomized, Open-label Study With Blinded Outcome Evaluation to Evaluate the Effects of Systolic Blood Pressure Lowering to Different Targets (Less Than 130 mmHg vs. Less Than 140 mmHg) on Diastolic Function Using Valsartan + Amlodipine in Patients With Hypertension and Diastolic Dysfunction
Brief Title: The Effects of Systolic Blood Pressure Lowering on Diastolic Function Using Valsartan + Amlodipine in Patients With Hypertension and Diastolic Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVAA489AUS01
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Results first posted 2011-03-10 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Hypertension; Diastolic Dysfunction
Keywords: Hypertension; systolic blood pressure; diastolic dysfunction; valsartan; amlodipine
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment regimen (Experimental): (Valsartan + Amlodipine to target SBP of < 140 mmHg)
  Interventions: Drug: valsartan; Drug: amlodipine
- Intensive treatment regimen (Experimental): (Valsartan + Amlodipine to target SBP < 130 mm Hg)
  Interventions: Drug: valsartan; Drug: amlodipine

INTERVENTIONS:
Drug: valsartan — 160 mg or 320 mg tablets once a day
  Other Names: Diovan
Drug: amlodipine — 5 mg or 10 mg tablets once a day
  Other Names: Norvasc

SUMMARY:
The purpose of this study is to determine the effects of treatment with valsartan + amlodipine to a target systolic blood pressure (SBP)<130 mmHg compared to the Joint National Commission on the Treatment of Hypertension 7 recommended target SBP of <140 mmHg on the intrinsic diastolic properties of the myocardium in patients with hypertension and echocardiographic evidence of diastolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 years or older
* Male and female patients are eligible. Female patients must be post-menopausal for one year, surgically sterile, or using effective contraceptive methods such as a double barrier method with spermicide, an intra-uterine device, or hormonal contraceptives. Post-menopausal women on a stable dose of hormone replacement therapy (HRT) for at least three (3) months prior to the screening visit are eligible for the study.
* Uncontrolled systolic hypertension on a maximum of two (2) antihypertensive medications at the time of screening.
* Echocardiographic ejection fraction ≥50% and evidence of diastolic dysfunction.
* Provide written informed consent to participate in the study prior to any screening or study procedures
* Have the ability to communicate well and comply with all study requirements

Exclusion Criteria:

* Severe hypertension defined as a MSSBP >200 mmHg and/or MSDBP >120 mmHg.
* History of a secondary cause of hypertension including but not limited to: coarctation of the aorta, hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's disease, pheochromocytoma, polycystic kidney disease, etc.
* Ejection fraction <50 %
* History of stroke, transient ischemic attack, myocardial infarction, coronary artery bypass graft surgery, or unstable angina pectoris within 6 months of screening
* Presence of clinically significant ventricular or supraventricular arrhythmias (e.g. atrial fibrillation/flutter)
* History of congestive heart failure
* History of diabetes mellitus
* History of renal impairment with serum creatinine >2.0 mg/dL at screening, history of dialysis, or history of nephritic syndrome
* Antihypertensive therapy with three (3) or more medications at the time of screening
* Active and/or treated malignancy of any organ system within twelve (12) months of enrollment, with the exception of localized basal cell carcinoma of the skin
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>5 mIU/ml)
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/m or 6 weeks post surgical bilateral oophorectomy with or without hysterectomy OR are using one or more of the following acceptable methods of contraception: barrier method with spermicidal agent, an intrauterine device, hormonal contraceptives, or total abstinence at the discretion of the investigator in cases where the age, career, lifestyle, or sexual orientation of the patient ensures compliance. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Reliable contraception should be maintained throughout the study
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of any drug including, but not limited to, any of the following: history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, bowel resection, gastric bypass, gastric stapling, or gastric banding, currently active, or active inflammatory bowel syndrome within 12 months prior to Visit 1, currently active gastritis, ulcers, or gastrointestinal/rectal bleeding, or urinary tract obstruction regarded as clinically meaningful by the investigator
* Pancreatic injury, pancreatitis or evidence of impaired pancreatic function/injury within 12 months prior to Visit 1
* Any serum AST or ALT elevation two (2) times the upper limit of normal

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Sites, USA, New Jersey, United States

REFERENCES:
- [Result] Solomon SD, Verma A, Desai A, Hassanein A, Izzo J, Oparil S, Lacourciere Y, Lee J, Seifu Y, Hilkert RJ, Rocha R, Pitt B; Exforge Intensive Control of Hypertension to Evaluate Efficacy in Diastolic Dysfunction Investigators. Effect of intensive versus standard blood pressure lowering on diastolic function in patients with uncontrolled hypertension and diastolic dysfunction. Hypertension. 2010 Feb;55(2):241-8. doi: 10.1161/HYPERTENSIONAHA.109.138529. Epub 2009 Dec 7. PMID 19996069

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive Treatment Regimen: (Valsartan + Amlodipine to target SBP < 130 mm Hg). Patients in the intensive treatment regimen had the study medication force-titrated to the maximum tolerated dose with the goal to achieve an SBP < 130 mm Hg.
  At week 0 patients received valsartan 160 mg + amlodipine 5 mg. At week 2, patients were force-titrated to valsartan 160 mg + amlodipine 10 mg. At week 4, patients were force titrated to valsartan 320 mg + amlodipine 10 mg. At week 8, patients who reached the SBP target < 130 mm Hg stayed on their current dose valsartan 320 mg + amlodipine 10 mg or the maximum tolerated dose as per the investigator's discretion. Patients not at SBP target < 130 mm Hg at week 8 or any study visits thereafter received other additional antihypertensive medications.
- Standard Treatment Regimen: (Valsartan + Amlodipine to target SBP of < 140 mmHg). Patients in the standard treatment regimen had the study medication up-titrated until the SBP goal of < 140 mm Hg was achieved.
  At week 0 patients received valsartan 160 mg + amlodipine 5 mg. At week 2 patients were up-titrated to valsartan 160 mg + amlodipine 10 mg only if they were not at SBP target < 140 mm Hg. At week 4 patients were up-titrated to valsartan 320 mg + amlodipine 10 mg only if they were not at SBP target < 140 mm Hg. Patients not at SBP target < 140 mm Hg by Week 8 or at any study visit thereafter received additional antihypertensive medications.
Period: Overall Study
Arm/Group | Intensive Treatment Regimen | Standard Treatment Regimen
Started | 114 | 115
Completed | 95 | 99
Not Completed | 19 | 16
Not completed — Adverse Event | 6 | 3
Not completed — Unsatisfactory therapeutic effect | 0 | 1
Not completed — Protocol Deviation | 3 | 1
Not completed — Patient withdrew consent | 7 | 6
Not completed — Lost to Follow-up | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Treatment Regimen | Standard Treatment Regimen | Total
Number analyzed (Participants) | 114 | 114 | 228
Age Continuous [Mean (Standard Deviation); unit: years] — In this study, even though the number of patients randomized to the intensive and standard treatment regimen were 114 and 115 respectively, analysis of the Baseline Measures was performed using the Safety Population. The Safety Population included all randomized patients who received at least one dose of study medication (Number of patients= 114 in both the treatment arms).
  years | 60.2 (10.03) | 58.9 (9.45) | 59.6 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants] — In this study, even though the number of patients randomized to the intensive and standard treatment regimen were 114 and 115 respectively, analysis of the Baseline Measures was performed using the Safety Population. The Safety Population included all randomized patients who received at least one dose of study medication (Number of patients= 114 in both the treatment arms).
  Participants
    Female | 61 | 54 | 115
    Male | 53 | 60 | 113

OUTCOME MEASURES:

1. Primary Outcome: Change in Lateral Mitral Annular Myocardial Relaxation Velocity
Description: Change from baseline in lateral mitral annular myocardial relaxation velocity (E') at Week 24
Time Frame: Baseline to 24 weeks after treatment
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Intensive Treatment Regimen | Standard Treatment Regimen
Number analyzed (Participants) | 98 | 98
cm/s | 1.544 (1.3946) | 1.476 (1.5985)

2. Secondary Outcome: Change in Left Atrial Size
Description: Change from baseline in left atrial size at Week 24
Time Frame: Baseline to 24 weeks after treatment
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intensive Treatment Regimen | Standard Treatment Regimen
Number analyzed (Participants) | 98 | 98
cm | -0.127 (0.3082) | -0.104 (0.2845)

3. Secondary Outcome: Change in Ratio of Peak E Wave Velocity/Lateral Mitral Annular Myocardial Relaxation Velocity
Description: Change from baseline in peak E-wave velocity / lateral mitral annular myocardial relaxation velocity (E/E') at Week 24
Time Frame: Baseline to 24 weeks after treatment
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Intensive Treatment Regimen | Standard Treatment Regimen
Number analyzed (Participants) | 98 | 98
ratio | -0.951 (2.1729) | -0.680 (2.0714)

4. Secondary Outcome: Percent Change From Baseline in Vascular Stiffness
Description: Percent change from baseline in Vascular Stiffness (measured by radial augmentation index [AI]) at Weeks 8 and 24
Time Frame: Baseline to 8 and 24 weeks after treatment
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: percentage of change in mean AI
Arm/Group | Intensive Treatment Regimen | Standard Treatment Regimen
Number analyzed (Participants) | 98 | 98
percentage of change in mean AI
  Week 8 | -7.89 (9.645) | -7.32 (11.970)
  Week 24 | -6.07 (10.582) | -5.63 (11.367)

5. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP)
Description: Change from baseline in msSBP at Weeks 8 and 24
Time Frame: Baseline to 8 and 24 weeks after treatment
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Intensive Treatment Regimen | Standard Treatment Regimen
Number analyzed (Participants) | 98 | 98
mm Hg
  Week 8 | -25.74 (16.112) | -22.31 (16.014)
  Week 24 | -30.37 (18.745) | -25.06 (17.074)

6. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: Change from baseline in msDBP at Weeks 8 and 24
Time Frame: Baseline to 8 and 24 weeks after treatment
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Intensive Treatment Regimen | Standard Treatment Regimen
Number analyzed (Participants) | 98 | 98
mm Hg
  Week 8 | -12.77 (10.118) | -12.62 (10.475)
  Week 24 | -15.21 (10.147) | -14.08 (11.163)

7. Secondary Outcome: Change in Estimated Central Aortic Pressure
Description: Change from baseline in estimated central aortic pressure at Weeks 8 and 24
Time Frame: Baseline to 8 and 24 weeks after treatment
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Intensive Treatment Regimen | Standard Treatment Regimen
Number analyzed (Participants) | 98 | 98
mm Hg
  Week 8 | -16.30 (12.483) | -14.68 (12.751)
  Week 24 | -17.71 (14.635) | -14.76 (12.689)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Even though the number of patients randomized to the intensive and standard treatment regimen were 114 and 115 respectively, analysis of the adverse events was performed in the Safety Population. The Safety Population included all randomized patients who received at least one dose of study medication (Number of patients= 114 in both treatment arms)
Arm/Group | Intensive Treatment Regimen | Standard Treatment Regimen
Serious Adverse Events (participants affected / at risk) | 3/114 | 3/114
Other Adverse Events (participants affected / at risk) | 49/114 | 41/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intensive Treatment Regimen (N=114) | Standard Treatment Regimen (N=114)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Appendicitis perforated (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intensive Treatment Regimen (N=114) | Standard Treatment Regimen (N=114)
Fatigue (General disorders) | 12 | 7
Oedema peripheral (General disorders) | 24 | 20
Upper respiratory tract infection (Infections and infestations) | 8 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 4
Dizziness (Nervous system disorders) | 16 | 9
Headache (Nervous system disorders) | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.